CLINICAL TRIAL: NCT02920398
Title: This Trial is Conducted in Europe and the United States of America. The Aim of This Trial is to Investigate Single Dose Pharmacokinetics (the Exposure of the Trial Drug in the Body) and Safety of Turoctocog Alfa Pegol From the Pivotal Process and Turoctocog Alfa Pegol From the Commercial Process in Patients With Severe Haemophilia A.
Brief Title: A Multi-centre, Comparative, Double Blind, Randomised Cross-over Trial Investigating Single Dose Pharmacokinetics and Safety of Turoctocog Alfa Pegol From the Pivotal Process and Turoctocog Alfa Pegol From the Commercial Process in Patients With Severe Haemophilia A
Acronym: pathfinder™7
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN7088-4033; 2015-005327-63 (EudraCT Number); U1111-1176-9253 (Other: WHO)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N8-GP pivotal (Experimental)
  Interventions: Drug: turoctocog alfa pegol
- N8-GP commercial (Active Comparator)
  Interventions: Drug: turoctocog alfa pegol

INTERVENTIONS:
Drug: turoctocog alfa pegol — Administered as intravenous injections at a dose of 50 U/kg. Patients will receive each product in a randomised cross-over design for comparison of the pharmacokinetics between turoctocog alfa pegol from the pivotal process and turoctocog alfa pegol from the commercial process.

SUMMARY:
Investigating single dose pharmacokinetics and safety of turoctocog alfa pegol from the pivotal process and turoctocog alfa pegol from the commercial process in patients with severe haemophilia A

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Ongoing participation in pathfinder™2
* Male, age at least 12 years at the time of signing informed consent (in certain countries the lower age limit will be 18 years, according to local requirements)

Exclusion Criteria:

* FVIII inhibitors (≥0.6 BU) at last visit in pathfinder™2 prior to entry in pathfinder™7
* Planned surgery during the trial
* Major surgery performed within 4 weeks prior to screening
* Previous participation in this trial. Participation is defined as signed informed consent
* Any disorder, except for conditions associated with haemophilia A, which in the investigator's opinion might jeopardise patient's safety or compliance with the protocol

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Area under the FVIII activity-time curve | From 0 to 96 hours post injection

SECONDARY OUTCOMES:
FVIII activity 30 min post administration - dose normalised to 50 U/kg | From time of trial product administration to 96 hours post-dose
Area under the FVIII activity-time curve from 0 to infinity | From time of trial product administration to 96 hours post-dose
Clearance in blood plasma of FVIII activity | From time of trial product administration to 96 hours post-dose
Incremental recovery in blood plasma of FVIII activity | From time of trial product administration to 96 hours post-dose
Terminal half-life | From time of trial product administration to 96 hours post-dose

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Nashville, Tennessee
- Novo Nordisk Investigational Site, Århus N, Denmark
- France (2):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Nantes
- Germany (3):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Frankfurt/M.
  - Novo Nordisk Investigational Site, Homburg
- Novo Nordisk Investigational Site, Groningen, Netherlands
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga